CLINICAL TRIAL: NCT00649714
Title: Single-Dose Food In Vivo Bioequivalence Study of Zonisamide Capsules (100 mg; Mylan) to Zonegran® Capsules (100 mg; Elan) in Healthy Volunteers
Brief Title: Fed Study of Zonisamide Capsules 100 mg and Zonegran® Capsules 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullivan, Global Head of Product Risk and Safety Management, Mylan, Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ZONI-0375
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Zonisamide

ARMS (2):
- 1 (Experimental): Zonisamide Capsules 100 mg
  Interventions: Drug: Zonisamide Capsules 100 mg
- 2 (Active Comparator): Zonegran® Capsules 100 mg
  Interventions: Drug: Zonegran® Capsules 100 mg

INTERVENTIONS:
Drug: Zonisamide Capsules 100 mg — 100mg, single dose fed
  Arms: 1
Drug: Zonegran® Capsules 100 mg — 100mg, single dose fed
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's zonisamide, 100 mg capsules to Elan's Zonegran® 100 mg capsules following a single, oral 100 mg (1 x 100 mg) dose administered under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years and older.
2. Sex: Male.
3. Weight: At least 60 kg (132 lbs) and within 15% of Ideal Body Weight (IBW), as referenced by the Table of ""Desirable Weights of Adults"" Metropolitan Life Insurance Company, 1999 (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
4. All subjects should be judged normal and healthy during a pre-study medical evaluation (physical examination, laboratory evaluation, hepatitis B and hepatitis C tests, HIV test, 12-lead ECG, and urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiate screen, phencyclidine, and methadone) performed within 14 days of the initial dose of study medication.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   1. Use of any tobacco products within 1 year of the start of the study.
   2. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.
   3. Ingestion of any vitamins or herbal products within the 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. A positive test for any drug included in the urine drug screen.
   6. History of drug and/or alcohol abuse.
3. Medications:

   1. Use of any prescription or over-the-counter (OTC) medications within the 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic disease.
   2. Acute illness at the time of either the pre-study medical evaluation or dosing.
   3. A positive HIV, hepatitis B, or hepatitis C test.
5. Abnormal and clinically significant laboratory test results:

   1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
   2. Abnormal and clinically relevant ECG tracing.
6. Donation or loss of a significant volume of blood or plasma (> 450 mL) within 28 days prior to the initial dose of study medication.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Allergy or hypersensitivity to zonisamide or any other sulfa drugs.
9. History of difficulties in swallowing, or any gastrointestinal disease which could affect the drug absorption.
10. Consumption of grapefruit or grapefruit containing products within 7 days of drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-12; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html